CLINICAL TRIAL: NCT01758172
Title: Comparison of Hemodynamic and Clinical Effects of Two Colloid Therapies in Post-operative Patients Undergoing Pancreaticoduodenectomy
Brief Title: Comparison of Hemodynamic Effects of Two Colloid Therapies in Post-operative Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Song Cheol Kim, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2008-1001
Record Dates: First submitted 2012-11-16; First posted 2013-01-01 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Pancreaticoduodenectomy
Keywords: pancreaticoduodenectomy; postoperative patient; colloid; albumin; hetastarch
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin (Active Comparator): albumin was administered to reach CVP up to 7mmHg
  Interventions: Drug: Albumin
- 6% hydroxyethyl starch 130/0.4 (Experimental): 6% hydroxyethyl starch 130/0.4 was administered to reach CVP up to 7mmHg
  Interventions: Drug: 6% hydroxyethyl starch 130/0.4

INTERVENTIONS:
Drug: 6% hydroxyethyl starch 130/0.4
  Arms: 6% hydroxyethyl starch 130/0.4
Drug: Albumin
  Arms: Albumin

SUMMARY:
From postoperative patients having undergone pancreaticoduodenectomy;

1. To compare the hemodynamic parameters from the patient administrated 5% HA and 6% Voluven
2. To assess the efficacy of the treatment as regards the clinical outcomes and laboratory parameters of the patient
3. To compare the safety of the 2 intravenous colloids in the patient population

ELIGIBILITY:
Inclusion Criteria:

* Subjects should be meet inclusion criteria to participated into the study

  1. Age-from 18-75 years adult
  2. In the immediate post-operative period of pancreaticoduodenectomy
  3. Written informed consent and admitted ICU immediate post-operative patient

Exclusion Criteria:

* Any patient meeting one or more of the following exclusion criteria may not be entered into the study.

  1. Refusal to participate in the study
  2. Evidence of pre-operative oliguria (Serum creatinine>1.5mmol/dL)
  3. Known Severe congestive heart failure (NYHAIII,IV)
  4. Known severe respiratory diseases (PaO2/FiO2 <200)
  5. Known coagulopathy (Platelet<100k/mm3, aPTT>70s, PT(INR)>2.5)
  6. Known allergy to hydroxyethyl starch
  7. Known pregnancy or lactation
  8. Has participated in any other clinical trial within 3months
  9. Any contraindication to Voluven® or albumin according to their package inserts.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure | post-op 24hr

SECONDARY OUTCOMES:
Volume(ml) of colloid | post-op 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: Song-cheol Kim, MD., PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea